CLINICAL TRIAL: NCT00349505
Title: Phase II Study of Intra-Peritoneal Hyper-Thermic Chemotherapy as Consolidation Therapy for Advanced Epithelial Ovarian Carcinoma
Brief Title: Intraperitoneal Hyperthermic Chemotherapy in Epithelial Ovarian Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHIPOVAC1; CSET 1058
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-09

CONDITIONS: Epithelial Ovarian Carcinoma; Figo Stage IIIC
Keywords: previous treatment surgery + 6 cycles of platinum based chemotherapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Procedure: hyper thermic chemo + surgery

SUMMARY:
Phase II to study results and morbidity of intra peritoneal hyper-thermic chemotherapy as consolidation therapy in patients with FIGO stage IIIC epithelial ovarian carcinoma treated by surgery and a total of 6 cycles of platinum based chemotherapy.

A second look operation is performed after treatment; during this second look secondary cytoreductive surgery is accepted without bowel resection.If none or milimetric peritoneal disease is obseved an intraperitoneal chemotherapy is achieve

ELIGIBILITY:
Inclusion Criteria:

epithelial ovarian carcinoma previous surgery + 6 cycles platinum based chemotherapy

-

Exclusion Criteria:

* Patients ASA 3 patients with no residual tumor at first operation negative microscopic second look

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Dominique ELIAS, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France